CLINICAL TRIAL: NCT05827952
Title: The Effect of Self-efficacy and Relationship Through Behavior Modification by Hybrid Mode in Caregivers With Toddler Receiving Early Intervention
Brief Title: The Effect of Self-efficacy and Relationship Through Behavior Modification by Hybrid Mode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-JIRB N202212060
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Caregivers With Toddler Receiving Early Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Groups/Cohorts (No Intervention): The "Self-learning group" was designed to provide a description of the goals of the course and a reading of the Atomic Habits book. In the first session, the goals of the study were explained, the basic abilities of the caregiver and the case, the games, the relationship, the main problems that the caregiver wanted to change, the "Parent Problem Checklist" to help assess the caregiver's direction in identifying their own expectations, and the caregiver's perceived barriers and difficulties. The next 8 weeks of the course are based on the parents' self-study progress, and the study provides an online platform or a paper sheet to keep track of the self-study process and to contact the researcher at any time if there are any unexpected situations or problems. The record sheets were returned at the end of the 8-week period, and the self-study group received a face-to-face consultation at the end of the post-test.
- Interventions (Experimental): Hybrid group used Atomic Habits (20-minute audiobook format), a role structure and a game structure, online schedule reminders more than twice a week and individual counseling sessions (online and physical) for one to two total interventions. The online schedule reminders consisted of four major habits, each with four concepts, to adapt the online audiobook interventions to the caregivers' relationship-building habits with the children A total of 16 sessions are delivered. Parents simply receive the course through digital media and complete the online schedule reminder within the course progress, narrowing down the indicators of habit change and achieving behavioral change through multiple executions.
  Interventions: Behavioral: behavior modification-Atomic Habit by hybrid

INTERVENTIONS:
Behavioral: behavior modification-Atomic Habit by hybrid — Atomic Habits (20-minute audiobook format), a role structure, and a game structure, online schedule reminders more than twice a week, and individual counseling sessions (online and physical) with one to two total interventions. The content of the online schedule reminders consisted of a total of four concepts for each of the four major habits, and a total of 16 sessions of the online audiobook interventions were adapted for the caregivers' relationship-building habits with the children.
  Arms: Interventions

SUMMARY:
The past literature supports the use of digital media as a medium to provide ongoing interventions for families caring for children with difficulties and the opportunity to intervene directly through caregivers, and to combine the advantages of hybrid physical and online interventions, applying different modes of teaching and interacting, satisfying the need for high frequency supervision and feedback for habit building, responding to difficulties and adjusting settings appropriately and immediately, in addition to providing timely assistance, by In addition to providing timely assistance, by changing parents' behavioral patterns and skills, it can increase the caregiver's level of implementation, thus establishing subtle changes and learning in daily life, promoting the quality of interaction and relationship building, and therefore providing intervention.

The study aims to use the new specific model of behavior modification-"Atomic Habit" as the basis for behavior change intervention, combining parental self-identification and children's play participation to establish good thinking and behavior patterns of caregivers, to increase self-identification and reduce stress, and to improve relationships and reduce conflict.

DETAILED DESCRIPTION:
Background: The COVID-19 pandemic had reduced access to early care, education, and life participation for families of children with developmental delay, resulting in deterioration of parental mental health, child deterioration, and parental unemployment. The literature supports that face-to-face or online caregiver-mediated interventions could promote child development, self-efficacy and reduce parental stress. The clinical practice of early care center in our hospital lacked a multi-disciplinary integrated relationship facilitation program for caregivers of children with developmental delay.

Purpose: The purpose of this study is to investigate the effects and examine of the behavior modification by hybrid in Stress, self-efficacy, relationships and conflict for caregivers Method: Caregivers of development delay children were recruited and randomly assigned to "Hybrid group"(n=20), and " Self-learning group" (n=19). After 8-weeks training (Online sessions and individual consultation sessions), the performance was assessed by a blinded assessor. The outcome measures included Intervention Fidelity, Parenting Sense of Confidence, Parenting Stress Index: Short form, The Conflict Tactics Scales: Parent Version, habit schedule record, satisfaction questionnaire.

Date analyzing: Collected data will be analyzed with Mann-Whinney U test, the Wilcoxon Signed Ranked Test, and Spearman correlation analysis by SPSS version 20.0, and alpha level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* children currently receiving care in early care;
* caregivers with a need to build parent-child relationships or improve self-efficacy;
* those who were able to use the pilot process and complete the homework, completing at least 10/12 training;
* those with internet access..

Exclusion Criteria:

* children currently receiving care in early care;
* caregivers with a need to build parent-child relationships or improve self-efficacy;
* those who were able to use the pilot process and complete the homework, completing at least 10/12 training;
* those with internet access.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Intervention Fidelity | through study completion, an average of 8 weeks
  A 4-point scale was used to understand parents' performance in knowledge, practice, participation, time, and use of resources in the implementation of the curriculum. The scale is "1" for totally disagree, "2" for somewhat agree, "3" for mostly agree, and "4 " indicates full agreement.
Parenting Sense of Confidence | Change from Baseline Parenting Sense of Confidence at 8 weeks
  By assessing parents' confidence and satisfaction with their role as a parent, 17 questions were asked on a 6-point scale ranging from "1" for strong agreement to "6" for strong disagreement, with higher scores indicating higher levels of parental confidence. The higher the score, the higher the parent's confidence. The scale is divided into two components, PSOC-E and PSOC-S, which reflect parental frustration, anxiety, and motivation, respectively, and the latter reflects competence, problem solving, and ability to perform the role of a parent. The Parental Effectiveness Scale (PSOC-E), which measures overall parental effectiveness, has a good internal reliability (Cronbach's alpha) of 0.76, while the Parental Satisfaction Scale (PSOC-S) has a good internal reliability (Cronbach's alpha) of 0.75; and can be used with caregivers of children of all ages.

SECONDARY OUTCOMES:
Parenting Stress Index: Short form | Change from Parenting Stress at 8 weeks
  The internal consistency of each subscale ranged from .856 to .908, and the total scale reached .947, representing a high level of consistency in the content of this scale.
The Conflict Tactics Scales: Parent Version | Change from Conflict Tactics Scales at 8 weeks
  The second part of the parent-child relationship was used to assess the parenting strategies used by parents/caregivers when children misbehaved, including "non-aggressive discipline" and "aggressive discipline".
Satisfaction Questionnaire: | through study completion, an average of 8 weeks
  A 12-question questionnaire was developed based on the course content, using a 4-point scale to collect information on caregivers' acceptance of the course, learning benefits, and to understand how caregivers feel they have changed.

CONTACTS AND LOCATIONS:
Overall Officials: FenLing Kuo, Master, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohan M, Bajaj G, Deshpande A, Anakkathil Anil M, Bhat JS. Child, Parent, and Play - An Insight into These Dimensions Among Children with and without Receptive Expressive Language Disorder Using Video-Based Analysis. Psychol Res Behav Manag. 2021 Jul 7;14:971-985. doi: 10.2147/PRBM.S306733. eCollection 2021. PMID 34262367
- [Background] Choo YY, Agarwal P, How CH, Yeleswarapu SP. Developmental delay: identification and management at primary care level. Singapore Med J. 2019 Mar;60(3):119-123. doi: 10.11622/smedj.2019025. PMID 30997518
- [Background] Corona LL, Stainbrook JA, Simcoe K, Wagner L, Fowler B, Weitlauf AS, Juarez AP, Warren Z. Utilization of telemedicine to support caregivers of young children with ASD and their Part C service providers: a comparison of intervention outcomes across three models of service delivery. J Neurodev Disord. 2021 Sep 15;13(1):38. doi: 10.1186/s11689-021-09387-w. PMID 34525940
- [Background] Edmondson D, Conroy D, Romero-Canyas R, Tanenbaum M, Czajkowski S. Climate change, behavior change and health: a multidisciplinary, translational and multilevel perspective. Transl Behav Med. 2022 May 25;12(4):503-515. doi: 10.1093/tbm/ibac030. PMID 35613001
- [Background] Hao Y, Franco JH, Sundarrajan M, Chen Y. A Pilot Study Comparing Tele-therapy and In-Person Therapy: Perspectives from Parent-Mediated Intervention for Children with Autism Spectrum Disorders. J Autism Dev Disord. 2021 Jan;51(1):129-143. doi: 10.1007/s10803-020-04439-x. PMID 32377905
- [Background] Hemdi A, Daley D. The Effectiveness of a Psychoeducation Intervention delivered via WhatsApp for mothers of children with Autism Spectrum Disorder (ASD) in the Kingdom of Saudi Arabia: A randomized controlled trial. Child Care Health Dev. 2017 Nov;43(6):933-941. doi: 10.1111/cch.12520. Epub 2017 Sep 20. PMID 28929582
- [Background] Humphries T, Kushalnagar P, Mathur G, Napoli DJ, Rathmann C, Smith S. Support for parents of deaf children: Common questions and informed, evidence-based answers. Int J Pediatr Otorhinolaryngol. 2019 Mar;118:134-142. doi: 10.1016/j.ijporl.2018.12.036. Epub 2018 Dec 29. PMID 30623850
- [Background] Ibanez LV, Kobak K, Swanson A, Wallace L, Warren Z, Stone WL. Enhancing interactions during daily routines: A randomized controlled trial of a web-based tutorial for parents of young children with ASD. Autism Res. 2018 Apr;11(4):667-678. doi: 10.1002/aur.1919. Epub 2018 Jan 7. PMID 29316336
- [Background] Klein CB, Swain DM, Vibert B, Clark-Whitney E, Lemelman AR, Giordano JA, Winter J, Kim SH. Implementation of Video Feedback Within a Community Based Naturalistic Developmental Behavioral Intervention Program for Toddlers With ASD: Pilot Study. Front Psychiatry. 2021 Dec 2;12:763367. doi: 10.3389/fpsyt.2021.763367. eCollection 2021. PMID 34925094
- [Background] Leadbitter K, Aldred C, McConachie H, Le Couteur A, Kapadia D, Charman T, Macdonald W, Salomone E, Emsley R, Green J; PACT Consortium. The Autism Family Experience Questionnaire (AFEQ): An Ecologically-Valid, Parent-Nominated Measure of Family Experience, Quality of Life and Prioritised Outcomes for Early Intervention. J Autism Dev Disord. 2018 Apr;48(4):1052-1062. doi: 10.1007/s10803-017-3350-7. PMID 29150738
- [Background] Li F, Wu D, Ren F, Shen L, Xue M, Yu J, Zhang L, Tang Y, Liu X, Tao M, Zhou L, Jiang L, Xu M, Li F. Effectiveness of Online-Delivered Project ImPACT for Children With ASD and Their Parents: A Pilot Study During the COVID-19 Pandemic. Front Psychiatry. 2022 Mar 24;13:806149. doi: 10.3389/fpsyt.2022.806149. eCollection 2022. PMID 35401276
- [Background] List JA, Pernaudet J, Suskind DL. Shifting parental beliefs about child development to foster parental investments and improve school readiness outcomes. Nat Commun. 2021 Oct 1;12(1):5765. doi: 10.1038/s41467-021-25964-y. PMID 34599167
- [Background] Luo J, Wang MC, Gao Y, Zeng H, Yang W, Chen W, Zhao S, Qi S. Refining the Parenting Stress Index-Short Form (PSI-SF) in Chinese Parents. Assessment. 2021 Mar;28(2):551-566. doi: 10.1177/1073191119847757. Epub 2019 May 9. PMID 31072108
- [Background] Waldman-Levi A, Bundy A, Shai D. Cognition Mediates Playfulness Development in Early Childhood: A Longitudinal Study of Typically Developing Children. Am J Occup Ther. 2022 Sep 1;76(5):7605205020. doi: 10.5014/ajot.2022.049120. PMID 35947034
- [Background] Wainer AL, Arnold ZE, Leonczyk C, Valluripalli Soorya L. Examining a stepped-care telehealth program for parents of young children with autism: a proof-of-concept trial. Mol Autism. 2021 May 8;12(1):32. doi: 10.1186/s13229-021-00443-9. PMID 33964979
- [Background] Salomone E, Pacione L, Shire S, Brown FL, Reichow B, Servili C. Development of the WHO Caregiver Skills Training Program for Developmental Disorders or Delays. Front Psychiatry. 2019 Nov 11;10:769. doi: 10.3389/fpsyt.2019.00769. eCollection 2019. PMID 31780960
- [Background] Salisbury MR, Roos LE, Horn SR, Peake SJ, Fisher PA. The Effectiveness of KEEP for Families of Children with Developmental Delays: Integrating FIND Video Coaching into Parent Management Training-Oregon Model: a Randomized Trial. Prev Sci. 2022 Aug;23(6):1029-1040. doi: 10.1007/s11121-022-01344-w. Epub 2022 Feb 2. PMID 35107694
- [Background] Sadeghi S, Pouretemad HR, Shalani B. Internet-based versus face-to-face intervention training for parents of young children with excessive screen-time and autism spectrum disorder-like symptoms: a comparative study. Int J Dev Disabil. 2021 Mar 8;68(5):744-755. doi: 10.1080/20473869.2021.1895699. eCollection 2022. PMID 36210895
- [Background] Ngai FW, Wong PW, Chung KF, Leung KY, Tarrant M. Randomized controlled trial of telephone-based cognitive-behavioral therapy on parenting self-efficacy and satisfaction. Transl Behav Med. 2019 Nov 25;9(6):1163-1168. doi: 10.1093/tbm/ibz017. PMID 30799485
- [Background] Neece CL, Chan N, Klein K, Roberts L, Fenning RM. Mindfulness-Based Stress Reduction for Parents of Children with Developmental Delays: Understanding the Experiences of Latino Families. Mindfulness (N Y). 2019 Jun;10(6):1017-1030. doi: 10.1007/s12671-018-1011-3. Epub 2018 Sep 6. PMID 31191735